CLINICAL TRIAL: NCT01917591
Title: Healing of Punch Graft Wounds With Two Biologic Exracellular Matrices; a Non-inferiority Study
Brief Title: Healing of Punch Graft Wounds. Comparative Study Between MariGen and Oasis: a Non-inferiority Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kerecis Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KS-0070
Record Dates: First submitted 2013-07-29; First posted 2013-08-06 (Estimated); Last update posted 2024-03-08 (Actual); Status verified 2017-02

CONDITIONS: Punch Biopsy Wounds; Healing Times
Keywords: Bandages; Biological Dressings; Chronic Disease; Collagen; Epithelium; Extracellular Matrix; Extra Cellular Matrix; Fibroblasts; Granulation Tissue; Leg Ulcer; Middle Aged; Prospective Studies; Soft Tissue Injuries; Treatment Outcome; Varicose Ulcer; Wound Healing; Wounds and Injuries; biopsy; autoimmunity
MeSH Terms: conditions — Chronic Disease; Leg Ulcer; Soft Tissue Injuries; Varicose Ulcer; Wounds and Injuries; Autoimmune Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MariGen Wound (Active Comparator): Fish derived extra cellular matrix
  Interventions: Device: Punch biopsies treated with MariGen Wound ECM dressing
- Oasis Sheet (Active Comparator): Pig intestine derived extra cellular matrix
  Interventions: Device: Punch biopsies treated with Oasis ECM dressing

INTERVENTIONS:
Device: Punch biopsies treated with MariGen Wound ECM dressing — Weekly dressing changes and review of wounds.
  Other Names: MariGen Wound ECM wound dressings.
  Arms: MariGen Wound
Device: Punch biopsies treated with Oasis ECM dressing — Weekly dressing changes and wound review
  Other Names: Oasis ECM wound dressing
  Arms: Oasis Sheet

SUMMARY:
The objective is to determine, if healing of punch biopsy wounds treated with the fish skin derived MariGen Wound dressing is non-inferior to healing with wounds treated with pig intestines derived Oasis Sheet wound dressing. Secondary endpoints are: Incidence of erythema, Pain, Infection, Quantitative measurements of autoantibodies at baseline and 4 weeks after start of treatment

ELIGIBILITY:
Inclusion Criteria:

* >18 yrs
* Healthy individual
* Signature of informed consent

Exclusion Criteria:

* Autoimmune disease
* Immunosuppressive treatment
* Use of addictive drugs
* Excessive use of alcohol
* Known fish allergy
* Known allergy to proteins with porcine origin
* Peripheral vascular disease
* Pregnant women
* Persons receiving anticoagulation therapy or systemic corticosteroids will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2013-01; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
wound healing | 28 days
  Time to epithelialisation

SECONDARY OUTCOMES:
Autoimmune investigations | 28 days
  Measurement of auto-antibodies including anti-collagen I and II antibodies
Incidence of erythema | 28 days
  Number of patients
Pain at wound site | 28 days
  number of patients with significant pain at wound site
Infection | 28 days
  Number of patients with infections

CONTACTS AND LOCATIONS:
Overall Officials: Hugrun Thorsteinsdottir, MD Derm, Principal Investigator — The National University Hospital of Iceland
Locations (1):
- Læknastofur Skipholti, Reykjavik, Iceland